CLINICAL TRIAL: NCT03977584
Title: Tau PET Longitudinal Substudy Associated With: A Double-Blind, Placebo-Controlled Parallel-Group Study in Preclinical PSEN1 E280A Mutation Carriers Randomized to Crenezumab or Placebo, and in Non-randomized, Placebo-treated Non-carriers From the Same Kindred, to Evaluate the Efficacy and Safety of Crenezumab in the Treatment of Autosomal-Dominant Alzheimer's Disease
Brief Title: Tau Positron Emission Tomography (PET) Longitudinal Substudy Associated With: Study of Crenezumab Versus Placebo in Preclinical Presenilin1 (PSEN1) E280A Mutation Carriers in the Treatment of Autosomal-Dominant Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Banner Alzheimer's Institute (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BN40199
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — crenezumab; (18F)GTP1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- [^18F]GTP1 in Mutation Carriers: Crenezumab (Experimental): Mutation-carrying participants receiving crenezumab in the main study NCT01998841 (GN28352) will receive up to three IV injections of [^18F]GTP1 and will undergo a tau PET scan after each IV injection of [^18F]GTP1.
  Interventions: Drug: Crenezumab; Other: [^18F]GTP1
- [^18F]GTP1 in Mutation Carriers: Placebo (Placebo Comparator): Mutation-carrying participants receiving placebo in the main study NCT01998841 (GN28352) will receive up to three IV injections of [^18F]GTP1 and will undergo a tau PET scan after each IV injection of [^18F]GTP1.
  Interventions: Drug: Placebo; Other: [^18F]GTP1
- [^18F]GTP1 in Non-carriers of Mutation: Placebo (Placebo Comparator): Non-carriers of the mutation receiving placebo in the main study NCT01998841 (GN28352) will receive up to three IV injections of [^18F]GTP1 and will undergo a tau PET scan after each IV injection of [^18F]GTP1.
  Interventions: Drug: Placebo; Other: [^18F]GTP1

INTERVENTIONS:
Drug: Crenezumab — Crenezumab will be administered subcutaneously (every 2 weeks) or IV (every 4 weeks) for at least 260 weeks.
  Other Names: MABT5102A
  Arms: [^18F]GTP1 in Mutation Carriers: Crenezumab
Drug: Placebo — Placebo matched to crenezumab will be administered subcutaneously (every 2 weeks) or IV (every 4 weeks) for at least 260 weeks.
  Arms: [^18F]GTP1 in Mutation Carriers: Placebo; [^18F]GTP1 in Non-carriers of Mutation: Placebo
Other: [^18F]GTP1 — IV [^18F]GTP1 will be administered up to three times. The first primary [^18F]GTP1 tau PET scan will occur during any visit in the main protocol NCT01998841 (GN28352) from Week 130 to Week 224 and the second [^18F]GTP1 tau PET scan from Week 248 to Week 260. The third and optional [^18F]GTP1 tau PET scan will supplement the two primary scans.

SUMMARY:
This substudy will evaluate the effect of crenezumab on the longitudinal tau burden in a subgroup of preclinical Presenilin1 (PSEN1) E280A mutation carriers and non-carriers, who were enrolled in study NCT01998841 (GN28352). Participants will receive up to three intravenous (IV) injections of [^18F] Genentech Tau Probe 1 (GTP1) and will undergo a tau positron emission tomography (PET) scan after each IV injection of [18^F]GTP1. The purpose of this substudy is to increase the understanding of disease progression in the preclinical stage of familial Alzheimer's Disease (AD).

ELIGIBILITY:
Inclusion Criteria:

- Enrolled in main Study NCT01998841 (GN28352).

Exclusion Criteria:

- Contraindication to PET scan procedures, possibly including, but not limited to current, past, or planned participation in studies involving radioactive agents, including the main Study NCT01998841 (GN28352) and this Tau PET substudy, such that the total research-related radiation dose to the participant in any given year would exceed the limits set forth in the U.S. Code of Federal Regulations (CFR) Title 21 Section 361.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Grupo Neurociencias de Antioquia, Medellín, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This sub-study enrolled participants from the main study: NCT01998841, who consented to participate in it. Participants took part in this sub-study from 10 Jun 2019 to 19 Apr 2022.
Pre-assignment Details: 114 participants enrolled in this sub-study.
Groups:
- Crenezumab - Mutation Carriers: Participants who were PSEN1 E280A mutation carriers and were administered crenezumab, 720 milligrams (mg), subcutaneously (SC), every two weeks (Q2W), or 60 milligrams per kilograms (mg/kg), intravenously (IV), every four weeks (Q4W) in the main study (NCT01998841) received up to three intravenous (IV) injections of [^18F] Genentech Tau Probe 1 (GTP1) and underwent a tau positron emission tomography (PET) scan after each IV injection of [^18F]GTP1.
- Placebo - Mutation Carriers: Participants who were PSEN1 E280A mutation carriers and were administered crenezumab matching placebo SC, Q2W or IV, Q4W in the main study (NCT01998841) received up to three IV injections of [^18F]GTP1 and underwent a tau PET scan after each IV injection of [^18F]GTP1.
- Placebo - Non-Carriers of Mutation: Participants who were non-carriers of PSEN1 E280A mutation and were administered crenezumab matching placebo SC, Q2W or IV, Q4W in the main study (NCT01998841) received up to three IV injections of [^18F]GTP1 and underwent a tau PET scan after each IV injection of [^18F]GTP1.
Period: Overall Study
Arm/Group | Crenezumab - Mutation Carriers | Placebo - Mutation Carriers | Placebo - Non-Carriers of Mutation
Started (114) | 44 | 39 | 31
Completed | 42 | 39 | 27
Not Completed | 2 | 0 | 4
Not completed — Reason not disclosed to prevent genetic unblinding | 2 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population (ITT) population included all randomized participants who received the assigned study treatment
Groups:
- Crenezumab - Mutation Carriers: Participants who were PSEN1 E280A mutation carriers and were administered crenezumab, 720 mg, SC, Q2W, or 60 mg/kg, IV, Q4W in the main study (NCT01998841) received up to three IV injections of [^18F]GTP1 and underwent a tau PET scan after each IV injection of [^18F]GTP1.
- Total: Total of all reporting groups
Arm/Group | Crenezumab - Mutation Carriers | Placebo - Mutation Carriers | Placebo - Non-Carriers of Mutation | Total
Number analyzed (Participants) | 44 | 39 | 31 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (5.5) | 36.7 (7.3) | 41.8 (8.0) | 37.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 29 | 23 | 73
  Male | 23 | 10 | 8 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 39 | 31 | 114
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 5 | 3 | 5 | 13
  Race: Asian | 0 | 0 | 0 | 0
  Race: Black or African American | 3 | 0 | 0 | 3
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: White | 17 | 22 | 14 | 53
  Race: Multiple | 15 | 8 | 12 | 35
  Race: Other | 4 | 6 | 0 | 10
  Race: Unknown | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Change in Tau Burden
Description: Tau is a protein that accumulates in Alzheimer's disease and damages brain cells including those essential for learning and memory. The effect of crenezumab on tau burden was assessed using [18F]GTP1 Tau PET. The annualized rate of change in tau burden from the first [18F]GTP1 scan of the standardized uptake ratio (SUVR) in the entorhinal cortex (Braak Stage 1) with an inferior cerebellum reference region was analyzed using a random coefficient regression model (RCRM). Braak staging classifies the degree of pathology in Alzheimer's disease. Braak stages 1 and 2 are used when neurofibrillary tangle involvement is confined mainly to the transentorhinal region of the brain, stages 3 and 4 when there is also involvement of limbic regions such as the hippocampus, and 5 and 6 when there is extensive neocortical involvement.
Time Frame: Baseline up to Week 149
Population: Modified Intent-to-Treat (mITT) population included all mutation carrier participants randomized in Study GN28352 (NCT01998841) and consented to the tau PET substudy who had received at least 1 dose of study drug.
Measure: Mean (Standard Error); unit: SUVR per year
Groups:
- Crenezumab - Mutation Carriers: Participants who were PSEN1 E280A mutation carriers and were administered crenezumab, 720 mg, SC, Q2W, or 60 mg/kg, IV, Q4W in the main study (NCT01998841) received up to three intravenous (IV) injections of [^18F]GTP1 and underwent a tau PET scan after each IV injection of [^18F]GTP1.
Arm/Group | Crenezumab - Mutation Carriers | Placebo - Mutation Carriers
Number analyzed (Participants) | 44 | 39
SUVR per year | 0.0124 (0.00752) | 0.0254 (0.00768)
Statistical Analysis 1: Comparison: Crenezumab - Mutation Carriers vs Placebo - Mutation Carriers; Analysis was based on RCRM using unstructured covariance matrix: GTP1 PET = Treatment * Analysis Year + Interactive Voice or Web Response System (IxRS) defined Age Group + IxRS defined Education History + IxRS defined apolipoprotein (APOE4) Carrier Status + IxRS defined Clinical Dementia Rating Global Score; Test type: Superiority; p = 0.1953, RCRM; Difference in Annualized Rate of Change = -0.0130, 95% CI 2-sided [-0.0327 to 0.0068], Standard Error of Mean 0.00993

ADVERSE EVENTS:
Time Frame: Up to Week 149
Description: Safety population included all participants randomized in Study GN28352 (NCT01998841) and consented to the tau PET substudy who had received at least 1 dose of study drug; participants were grouped according to the actual treatment received and the mutation status. Pooled data has been reported for the SAEs and non-serious AEs in order to maintain blinding of the participant's mutation status and treatment group.
Groups:
- Crenezumab - Mutation Carriers: Participants who were PSEN1 E280A mutation carriers and were administered crenezumab, 720 mg, SC, Q2W, or 60 mg/kg, IV, Q4W in the main study (NCT01998841) received up to three IV injections of [^18F] GTP1 and underwent a tau PET scan after each IV injection of [^18F]GTP1.
- Pooled Placebo: Carriers and non-carriers of PSEN1 E280A mutation who received matching placebo SC, Q2W or IV, Q4W in the main study (NCT01998841), received up to three IV injections of [^18F]GTP1 and underwent a tau PET scan after each IV injection of [^18F]GTP1.
- Combined Blinded: All participants who were carriers and non-carriers of PSEN1 E280A mutation and who received either crenezumab, 720 mg, SC, Q2W, or 60 mg/kg, IV, Q4W or matching placebo SC, Q2W or IV, Q4W in the main study (NCT01998841) received up to three IV injections of [^18F]GTP1 and underwent a tau PET scan after each IV injection of [^18F]GTP1.
Arm/Group | Crenezumab - Mutation Carriers | Pooled Placebo | Combined Blinded
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/70 | 0/114
Serious Adverse Events (participants affected / at risk) | 4/44 | 5/70 | 9/114
Other Adverse Events (participants affected / at risk) | 43/44 | 67/70 | 110/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Crenezumab - Mutation Carriers (N=44) | Pooled Placebo (N=70) | Combined Blinded (N=114)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions (General disorders) | 4 (5) | 5 (5) | 1 (1)
Infections and infestations (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0 (0) | 0/39 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crenezumab - Mutation Carriers (N=44) | Pooled Placebo (N=70) | Combined Blinded (N=114)
Infections and infestations (Infections and infestations) | 36 (67) | 54 (134) | 90 (201)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 22 (58) | 30 (70) | 52 (128)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 20 (30) | 28 (40) | 48 (70)
Nervous system disorders (Nervous system disorders) | 16 (32) | 26 (46) | 42 (78)
Psychiatric disorders (Psychiatric disorders) | 10 (17) | 22 (29) | 32 (46)
Gastrointestinal disorders (Gastrointestinal disorders) | 15 (22) | 15 (20) | 30 (42)
General disorders and administration site conditions (General disorders) | 6 (9) | 14 (16) | 20 (25)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 4 (5) | 14 (17) | 18 (22)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 6 (6) | 8 (10) | 14 (16)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 6 (8) | 8 (8) | 14 (16)
Renal and urinary disorders (Renal and urinary disorders) | 6 (6) | 7 (8) | 13 (14)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 8 (8) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03977584/Prot_SAP_000.pdf